CLINICAL TRIAL: NCT01519804
Title: A Randomized, Phase II, Multicenter, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Onartuzumab (Metmab) in Combination With Paclitaxel + Cisplatin or Carboplatin as First-Line Treatment for Patients With Stage IIIb (T4 Disease) or IV Squamous Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Study of Onartuzumab (MetMAb) Versus Placebo in Combination With Paclitaxel Plus Platinum in Patients With Squamous Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GO27820
Record Dates: First submitted 2011-12-19; First posted 2012-01-27 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Cisplatin; Carboplatin; onartuzumab; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- MetMAb+paclitaxel+platinum (Experimental)
  Interventions: Drug: cisplatin/carboplatin; Drug: onartuzumab; Drug: paclitaxel
- Placebo+paclitaxel+platinum (Active Comparator)
  Interventions: Drug: Placebo; Drug: cisplatin/carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: Placebo — Matching onartuzumab (MetMAb) placebo iv, Day 1 of each 21-day cycle
  Arms: Placebo+paclitaxel+platinum
Drug: cisplatin/carboplatin — standard dose iv, Day 1 of each 21-day cycle, 4 cycles
Drug: onartuzumab — 15 mg/kg iv, Day 1 of each 21-day cycle
  Other Names: MetMAb
  Arms: MetMAb+paclitaxel+platinum
Drug: paclitaxel — 200 mg/m2 iv, Day 1 of each 21-day cycle, 4 cycles

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled study will evaluate the efficacy and safety of onartuzumab (MetMAb) in combination with paclitaxel plus platinum in patients with incurable Stage IIIB or Stage IV squamous non-small cell lung cancer (NSCLC). Patients will be randomized to receive either onartuzumab (MetMAb) 15 mg/kg iv or placebo on Day 1 of each 21-day cycle in combination with 4 cycles of paclitaxel 200 mg/m2 iv and platinum (carboplatin/cisplatin) iv on Day 1 of each 21-day cycle. Patients who have not progressed after 4 cycles will continue with either onartuzumab (MetMAb) or placebo as maintenance therapy until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Histologically or cytologically confirmed Stage III B or Stage IV squamous non-small cell lung cancer (NSCLC)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* No prior chemotherapy for squamous NSCLC
* Adequate tissue for central IHC assay of Met receptor, and EGFR testing if EGFR status is unknown
* Radiographic evidence of disease

Exclusion Criteria:

* Prior systemic treatment for Stage IIIB or IV squamous NSCLC
* NSCLC with histology classified as adenocarcinoma, large cell, mixed adenosquamous, or NSCLC not otherwise specified (NOS)
* Prior exposure to experimental treatment targeting either the HGF or Met pathway
* Patients with tumors confirmed to have EGFR-activating mutations who are suitable for anti-EGFR therapy (e.g. gefitinib or erlotinib), as determined by the investigator
* Uncontrolled brain metastases and treatment by neurosurgical resection or brain biopsy within 4 weeks prior to Day 1 of Cycle 1
* History of another malignancy in the previous 3 years except for prior history of in situ cancer or basal or squamous cell skin cancer
* Pregnant or lactating women
* Uncontrolled diabetes
* Impaired bone marrow, liver or renal function as defined by protocol
* Significant history of cardiovascular disease
* Positive for HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2012-04; Primary Completion 2014-01 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (tumor assessments according to RECIST criteria) | up to approximately 32 months
Progression-free survival: Subgroup of patients with Met diagnostic-positive squamous NSCLC | up to approximately 32 months

SECONDARY OUTCOMES:
Overall survival | up to approximately 32 months
Overall response rate (tumor assessments according to RECIST criteria) | up to approximately 32 months
Duration of response (time from first documented objective response to disease progression) | up to approximately 32 months
Disease control rate (rate of partial response plus complete response plus stable disease for at least 6 weeks) | up to approximately 32 months
Safety: Incidence of adverse events | up to approximately 32 months
Pharmacokinetics: serum concentration (Cmin/Cmax) | Pre- and post-dose on Day 1 of Cycles 1, 2 and 4 and up to 2 years
Plasma concentrations of paclitaxel/platinum | Pre- and post-dose on Day 1 of Cycles 1 and 4
Serum levels of anti-therapeutic antibodies (MetMAb ATAs) | Pre-dose Day 1 of Cycles 1, 2 and 4

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (64):
- United States (31):
  - Huntsville, Alabama
  - Scottsdale, Arizona
  - Bakersfield, California
  - Fullerton, California
  - Los Angeles, California
  - Northridge, California
  - Sacramento, California
  - San Luis Obispo, California
  - Santa Barbara, California
  - Stanford, California
  - Grand Junction, Colorado
  - Boynton Beach, Florida
  - Orlando, Florida
  - Weston, Florida
  - Marietta, Georgia
  - Chicago, Illinois
  - Harvey, Illinois
  - Fort Wayne, Indiana
  - Indianapolis, Indiana
  - Muncie, Indiana
  - Metairie, Louisiana
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Hickory, North Carolina
  - Cleveland, Ohio
  - Middletown, Ohio
  - Bend, Oregon
  - Pittsburgh, Pennsylvania
  - Seattle, Washington
- Argentina (3):
  - Buenos Aires
  - La Rioja
  - Santa Rosa
- France (4):
  - Grenoble
  - Lyon
  - Paris
  - Rennes
- Germany (6):
  - Berlin
  - Göttingen
  - Halle
  - Immenhausen
  - München
  - Münster
- Israel (4):
  - Afula
  - Ashkelon
  - Tel Aviv
  - Ẕerifin
- Italy (5):
  - Avellino, Campania
  - Napoli, Campania
  - Udine, Friuli Venezia Giulia
  - Cremona, Lombardy
  - Milan, Lombardy
- Latvia (3):
  - Daugavpils
  - Liepāja
  - Riga
- Spain (4):
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Pamplona, Navarre
  - Zaragoza, Zaragoza
- United Kingdom (4):
  - Aberdeen
  - Birmingham
  - Bournemouth
  - Leeds